CLINICAL TRIAL: NCT01482975
Title: Tailored Interventions to Prevent Substance Abuse
Acronym: Project BEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rhode Island (Other)
Responsible Party: Principal Investigator, Wayne F. Velicer, Professor, University of Rhode Island
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: DA020112
Record Dates: First submitted 2011-11-29; First posted 2011-12-01 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Prevention Harmful Effects
Keywords: tobacco; alcohol; diet; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smoking and Alcohol Prevention (Experimental): TTM expert system
  Interventions: Other: Tailored computer based intervention
- Diet and Exercise (Active Comparator): TTM expert system
  Interventions: Other: Tailored computer intervention

INTERVENTIONS:
Other: Tailored computer based intervention — Best practices for TTM tailored communication with two types of feedback: normative - compared to peer and ipsative - self compared to previous assessment.
  Other Names: Tailored computer based interventions
  Arms: Smoking and Alcohol Prevention
Other: Tailored computer intervention — Best practices for TTM tailored communication with two types of feedback: normative - compared to peer and ipsative - self compared to previous assessment
  Arms: Diet and Exercise

SUMMARY:
The overarching objective of this research is to prevent substance use in early adolescents through the use of innovative interactive interventions tailored to each individual's particular risk profile for using cigarettes and alcohol. The specific aims are: (1) To test the effectiveness of the computer-based profile-based tailored interventions to keep early adolescents smoke-free compared to a comparison group; (2) To test the effectiveness of the computer-based profile-based tailored interventions to keep early adolescents from using alcohol compared to a comparison group; and (3) To replicate findings that the tailored diet and physical activity interventions will be effective in reducing these two high risk behaviors as part of the comparison condition.

DETAILED DESCRIPTION:
Research across age groups (elementary, middle and high school), populations (U.S., U.K., and Israel), and substances (tobacco, alcohol and other drugs) has consistently identified four clusters of non-users who vary in their risks for substance use: (1) Most Protected from substance use; (2) High Risk to use substances; (3) Ambivalent about staying substance free; and (4) Risk Denial about substance use. These profiles have demonstrated both internal and external validity as well as good ability to predict future substance use and, therefore, provide an opportunity to develop a new approach to prevention. These profiles will be employed as the basis for designing two innovative computer-based interventions to prevent substance abuse by adolescents. The two new tailored interventions (smoking prevention and alcohol prevention) will be developed and tested in a school-based clinical trial. The comparison group will receive two previously developed and tested tailored health behavior interventions (diet and physical activity).

ELIGIBILITY:
Inclusion Criteria:

* 6th grade student in one of 20 participating Middle Schools in RI
* English speaking
* Student Assent

Exclusion Criteria:

* Parent refusal for child to participate

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4158 (Actual)
Dates: Start 2007-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Smoking Prevention | 36 months
  Percent reporting being smoke-free at 36 months
Alcohol Use Prevention | 36 months
  Percent reporting being alcohol-free at 36 months
Exercise | 36 months
  Percentage of baseline at-risk participants who reach the Regular Exercise criteria (60 minutes a day/five days per week).
Diet | 36 months
  Percentage of at-risk participants at baseline who reach Diet Criteria (five or more a day servings of fruits and vegetables).

CONTACTS AND LOCATIONS:
Overall Officials: Wayne F Velicer, PhD, Principal Investigator — Univeristy of Rhode Island
Locations (1):
- University of Rhode Island, Kingston, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No